CLINICAL TRIAL: NCT02179723
Title: Clinical Study Into the Cosmetic Results of Leukosan Adhesive vs. Transcutaneous Wound Suture With Laparoscopic Trocar Incision
Brief Title: Clinical Study Into the Cosmetic Results of Leukosan Adhesive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Stephanie Krause (Industry)
Responsible Party: Sponsor-Investigator, Dr. Stephanie Krause, Scientific Affairs, Wound Care, BSN Medical GmbH
Organization: BSN Medical GmbH (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: BSNMedicalC09962; PV4003 (Other: Ethik Kommission der Aerztekammer Hamburg)
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Wound Healing Cosmetic Result
Keywords: wound healing; cosmetic results; trocar incision

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Leukosan Adhesive (Experimental): Leukosan Adhesive applied to one wound (left or right)
  Interventions: Device: Leukosan Adhesive; Device: Transcutaneous suture
- Transcutaneous suture (Active Comparator): Transcutaneous suture applied to second wound (left or right)
  Interventions: Device: Leukosan Adhesive; Device: Transcutaneous suture

INTERVENTIONS:
Device: Leukosan Adhesive — Leukosan adhesive applied to one wound
Device: Transcutaneous suture — Transcutaneous suture applied to one wound

SUMMARY:
This clinical study aims to assess whether the benefits of using Leukosan Adhesive on trocar incisions are greater or equivalent to those provided by the standard therapy of transcutaneous sutures.

In particular, it tests the long-term cosmetic result after 3 months, the safety and tolerance, as well as the practicality of treatment with Leuksan Adhesive.

An open, randomised, controlled, prospective, single location, clinical study of women of ages between 18 and 60 years within the time span of March 2013 and April 2013.

DETAILED DESCRIPTION:
The medical devices compared were EU (European Union) approved market-ready products with relevant designation according to the legal requirements for medical devices and according to Council guideline 93/42/EWG dated 14th July.

Leukosan Adhesive is a sterile, ultra high viscose adhesive for external skin closure. Due to the skin's moisture, this skin adhesive polymerizes within seconds into a flexible film firmly holding the edges of the wound together and protecting the wound itself.

Premilene DSMP 24, 3/8 needle, thread 3/0 denier was used a a comparison. This suture material was the standard suture material used in the study centre.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 60
* Undergone laparoscopic operation with 2 mirror image trocar incisions
* Willing to attend examination at clinic at 7-12 days and 10-14 weeks
* Signed agreement by participant

Exclusion Criteria:

* Length of laparoscopic operation more than 2 hours
* Hospitalisation due to complications
* Circumstances leading to difference in trocar incisions
* Existing scar less than 3 cm from the operation point
* Diabetic condition melitis HbA1c>9mg/d
* Known allergy to tissue adhesive
* Participation in another study within 30 days

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Patient's satisfaction with cosmetic appearance/result of the wound | 3 months post operation
  The primary outcome was the satisfaction of the patients with the cosmetic result of the wound healing after 3 months. This was measured by a visual analogue scale. In order to validate this result, an additional known wound assessment instrument, an ordinal scaled index, was implemented and the assessment of independent assessors was called on.

SECONDARY OUTCOMES:
The incidence of complication | 7-12 days post-operation
  7-12 days post-operation patients were examined for complications in treatment such as wound dehiscence, maceration, redness, overheating and pain
Intensity of pain | 7-12 days post-operation
  7-12 days post-operation patients were examined for intensity of pain
Investigator's assessment of cosmetic outcome | At 3 months post-operation
  The Investigator examined patients to assess the cosmetic outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Buchweitz, Priv.Doz., Principal Investigator — Tagesklinik Altonaer Strasse
Locations (1):
- Tagesklinik Altonaer Strasse, Hamburg, Germany

REFERENCES:
- [Background] Rosen DM, Carlton MA. Skin closure at laparoscopy. J Am Assoc Gynecol Laparosc. 1997 May;4(3):347-51. doi: 10.1016/s1074-3804(05)80226-9. PMID 9154784
- [Background] Matin SF. Prospective randomized trial of skin adhesive versus sutures for closure of 217 laparoscopic port-site incisions. J Am Coll Surg. 2003 Jun;196(6):845-53. doi: 10.1016/s1072-7515(03)00119-4. PMID 12788419
- [Background] Buchweitz O, Wulfing P, Kiesel L. A prospective randomized trial of closing laparoscopic trocar wounds by transcutaneous versus subcuticular suture or adhesive papertape. Surg Endosc. 2005 Jan;19(1):148-51. doi: 10.1007/s00464-004-9043-2. Epub 2004 Nov 18. PMID 15549624
- [Background] Chen K, Klapper AS, Voige H, Del Priore G. A randomized, controlled study comparing two standardized closure methods of laparoscopic port sites. JSLS. 2010 Jul-Sep;14(3):391-4. doi: 10.4293/108680810X12924466006729. PMID 21333194
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848
- [Derived] Buchweitz O, Frye C, Moeller CP, Nugent W, Krueger E, Nugent A, Biel P, Juergens S. Cosmetic outcome of skin adhesives versus transcutaneous sutures in laparoscopic port-site wounds: a prospective randomized controlled trial. Surg Endosc. 2016 Jun;30(6):2326-31. doi: 10.1007/s00464-015-4474-5. Epub 2015 Oct 1. PMID 26428200